CLINICAL TRIAL: NCT01763515
Title: The Effects of Laterally Wedged Insoles on Symptoms Reduction of Patients With Knee Osteoarthritis
Brief Title: Laterally Wedged Insoles for Patients With Knee Osteoarthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Farnaz Dehgan Hosseinabadi, Dr., Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13913008
Record Dates: First submitted 2012-12-28; First posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Joint Diseases; Arthritis; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Arthritis; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laterally wedged insoles (Experimental): Patients will use laterally wedged insoles with 5o tilt toward medial side and made of ethylene vinyl acetate coated with leather. The medial thickness is 4 mm with lateral thickness of 10 mm.
  Interventions: Procedure: Laterally wedged insoles

INTERVENTIONS:
Procedure: Laterally wedged insoles — Patients will use laterally wedged insoles with 5o tilt toward medial side and made of ethylene vinyl acetate coated with leather. The medial thickness is 4 mm with lateral thickness of 10 mm.

SUMMARY:
Knee osteoarthritis is a common problem with the disease prevalence increasing with advancing age. This study will be performed in the purpose of determination the effects of laterally wedged insoles on symptoms reduction of patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis is a common problem with the disease prevalence increasing with advancing age. Because of the high incidence of knee osteoarthritis in the elderly and the seriousness of drug effects in this age group and lack of controlled study in our country regarding the possible benefits or lack of benefit of laterally wedged insoles in patients with knee osteoarthritis and also due to strike, and results of mixed in other studies, this study will be performed in the purpose of determination the effects of laterally wedged insoles on symptoms reduction of patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic medial femorotibial knee OA,
* Daily knee pain for at least 1 month in the last 3 months,
* Radiographic evidence of medial femorotibial knee OA,
* Normal erythrocyte sedimentation rate.

Exclusion Criteria:

* Secondary knee OA, hip OA, symptomatic foot deformities, articular space loss more or the same as lateral femorotibial side in radiography,
* Knee joint lavage in past 3 months,
* Intra-articular corticosteroid injection during the past 3 months,
* Tibial osteotomy during last 5 years and changes in drug treatment for OA during last week.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-08 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in knee pain severity after 2 months. | Up to 2 months
  The pain score (100 mm Visual Analogue Score ) is evaluated at baseline and then after 2 months of therapy.

SECONDARY OUTCOMES:
Change from baseline in knee's functional degree after 2 months. | Up to 2 months.
  Knee's functional degree (Edinburg Index) is evaluated at baseline and then 2 months after therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Farnaz Dehghan, MD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Department of Rehabilitation, Alzahra Hospital, Isfahan, Isfahan, Iran

REFERENCES:
- [Background] Hinman RS, Bowles KA, Bennell KL. Laterally wedged insoles in knee osteoarthritis: do biomechanical effects decline after one month of wear? BMC Musculoskelet Disord. 2009 Nov 25;10:146. doi: 10.1186/1471-2474-10-146. PMID 19939281
- [Background] Bennell K, Bowles KA, Payne C, Cicuttini F, Osborne R, Harris A, Hinman R. Effects of laterally wedged insoles on symptoms and disease progression in medial knee osteoarthritis: a protocol for a randomised, double-blind, placebo controlled trial. BMC Musculoskelet Disord. 2007 Sep 24;8:96. doi: 10.1186/1471-2474-8-96. PMID 17892539
- [Background] Pham T, Maillefert JF, Hudry C, Kieffert P, Bourgeois P, Lechevalier D, Dougados M. Laterally elevated wedged insoles in the treatment of medial knee osteoarthritis. A two-year prospective randomized controlled study. Osteoarthritis Cartilage. 2004 Jan;12(1):46-55. doi: 10.1016/j.joca.2003.08.011. PMID 14697682